CLINICAL TRIAL: NCT06573333
Title: Effects of Timing of Cord Clamping on Serum Calcium Levels in Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Umair Anees Qureshi, Doctor, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 369452
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Serum Calcium Concentration

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trails
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15 seconds (Experimental): Umbilical Cord will be clamped after 15s of birth and Serum calcium levels will be measured at 6 hours of life
  Interventions: Procedure: Umblical Cord Clamping
- 30seconds (Experimental): Umbilical Cord will be clamped after 30s of birth and Serum calcium levels will be measured at 6 hours of life
  Interventions: Procedure: Umblical Cord Clamping
- 60seconds (Experimental): Umbilical Cord will be clamped after 60s of birth and Serum calcium levels will be measured at 6 hours of life
  Interventions: Procedure: Umblical Cord Clamping
- 120 seconds (Experimental): Umbilical Cord will be clamped after 120s of birth and Serum calcium levels will be measured at 6 hours of life
  Interventions: Procedure: Umblical Cord Clamping

INTERVENTIONS:
Procedure: Umblical Cord Clamping — Umbilical Cord will be clamped using a plastic clamp at the noted time after delivery of the neonate

SUMMARY:
Title: Effect of timing of cord clamping of serum calcium levels in neonates Background: Hypocalcemia is a common metabolic problem in neonatal period. Most cases of hypocalcemia are asymptomatic however, the symptomatic cases require prompt management.

Objective: The objective is to determine the effects of early and delayed cord on serum calcium level in neonates Study Design: Randomized Controlled Trial

DETAILED DESCRIPTION:
Place and Duration of Study: PEMH Rawalpindi and CMH Rawalpindi from January 2024 to July 2024.

Patients and Methods: Total sample size of 200 neonates will be included in the study divided into four groups with cord clamping at 15s, 30s, 60s, 120s each group will have a total of 50 neonates. Blood sampling for CBC / CRP / S. Electrolytes (Na, K, Total Ca, Ionized Ca, Mg), S Calcitonin, ABGs (HCO3 Levels) samples will be collected at 6 hours of life.

* Inclusion Criteria: Neonates born at gestational age 37 weeks to 41 weeks with no maternal complication. Parents who give consent for inclusion in the study
* Exclusion Criteria: Mothers with evidence of clinical disease (diabetes, preeclampsia, hypertension). Babies with congenital malformations and intrauterine growth restriction.

Expected Results: Research data on serum Calcium levels in neonates have shown no correlation to timing of cord clamping. Same results are expected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at gestational age 37 weeks to 41 weeks with no maternal complication. Parents who give consent for inclusion in the study

Exclusion Criteria:

* Mothers with evidence of clinical disease (diabetes, preeclampsia, hypertension). Babies with congenital malformations and intrauterine growth restriction.

Ages: 1 Minute to 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Effects of Timing of Cord Clamping on Serum Calcium Levels in Neonates | at 6 hours of life
  Serum Calcium Levels

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Khushdil, MBBS, Principal Investigator — Military Hospital Rawalpindi
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan